CLINICAL TRIAL: NCT05906485
Title: Randomized Controlled Trials of the Effects of Near-infrared Spectroscopy (fNIRS) Neurofeedback Training Coupled With Virtual Reality Technology in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: fNIRS Neurofeedback Training Using Virtual Reality in Children With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kathy Shum, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA200247
Record Dates: First submitted 2023-05-22; First posted 2023-06-18 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: ADHD
Keywords: fNIRS Neurofeedback Training; Virtual Reality; Children with ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Experimental group: receives 8-week functional near-infrared spectroscopy (fNIRS) neurofeedback training (coupled with virtual reality) in Phase 1, twice per week, each lasts 1 hour.
  Active control group: receives 8-weeks computerized cognitive training in Phase 1, twice per week, each lasts 35 minutes.
  Waitlist control group: either receives 8-weeks fNIRS neurofeedback training (coupled with virtual reality) or computerized cognitive training in Phase 2 (i.e., after the completion of training for intervention group and active control group).
Who Masked: Participant
Masking Description: Participants will be randomly allocated into groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group: fNIRS Neurofeedback-VR Training Group (Experimental): The experimental group will receive 16 sessions of training, 1 hour each, conducted twice per week over a period of 8 weeks. A classroom setting will be stimulated using VR and participants will be asked to complete some academic-related tasks during the stimulated lessons. The sensor on the neurofeedback device worn by the participants will detect changes in the blood oxy-hemoglobin level in brain cortical tissue and feedback to the participants via visual images or auditory sounds from the computer. Through practice, participants will learn to manipulate their attention, presumably by altering brain activities.
  Interventions: Behavioral: fNIRS Neurofeedback-VR Training
- Active Control Group: Computerized Cognitive Training Group (Active Comparator): The computerized cognitive training group will receive 16 sessions of training, 35 minutes each, conducted twice per week over a period of 8 weeks. Participants will be asked to complete a set of computerized tasks using Cogmed, a digital training programme which is proven to enhance working memory and attention level in children.
  Interventions: Behavioral: Computerized Cognitive Training
- Waitlist Control Group (Other): The waitlist control group will not receive any intervention until the intervention arms complete their training. Depending on the availability, either the fNIRS Neurofeedback-VR Training or the Computerized Cognitive Training will be offered to this group.
  Interventions: Behavioral: fNIRS Neurofeedback-VR Training; Behavioral: Computerized Cognitive Training

INTERVENTIONS:
Behavioral: fNIRS Neurofeedback-VR Training — In the fNIRS Neurofeedback-VR Training, we have designed a classroom scenario modeled and children are expected to learn how to regulate their attention based on the feedback provided by the fNIRS on the oxygenated haemoglobin level in their prefrontal cortex.
  Arms: Experimental Group: fNIRS Neurofeedback-VR Training Group; Waitlist Control Group
Behavioral: Computerized Cognitive Training — In the Computerized Cognitive Training, children will complete a range of tasks covering attention control and working memory using a conventional training programme, namely Cogmed.
  Arms: Active Control Group: Computerized Cognitive Training Group; Waitlist Control Group

SUMMARY:
The study aims to explore the effectiveness of neurofeedback training on improving attention and inhibitory control of children with attention-deficit/hyperactivity disorder (ADHD) in Hong Kong. This study will contribute to the current understanding of the alternative treatments for ADHD, and hopefully help to mobilize more resources to support children with ADHD. The programme includes the following components:

Participants will be randomly assigned to the neurofeedback training group (with virtual reality [VR] technology applied), the computerized cognitive training group, or the waitlist control group. All participants will complete a total of 16 training sessions in 8 weeks (twice a week), and each session will last around 35 to 60 mins.

To investigate the intervention effectiveness, children will be asked to complete a set of cognitive tests covering inhibitory control, attention, and working memory prior to the intervention (i.e., Time 1), immediately after the 8-week training (i.e., Time 2), and 2 months after the training (i.e., Time 3, a 2-month follow up). The assessment will take around 1 hour and it will be conducted at the laboratory at the University of Hong Kong. Also, parents and teachers will be asked to complete a questionnaire assessing children's behaviours at home and schools at 3 timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7- 12
* Clinical diagnosis of ADHD
* Significant teacher- or parent-reported attention problems during screening

Exclusion Criteria:

* IQ under 70, as measured on Raven's Progressive Matrices
* Hearing, visual, or physical impairments that might hinder participation in the training and assessment activities
* Clinical diagnosis and suspected cases of Autism Spectrum Disorder (ASD)
* Prior or current participation in NFT
* Current participation in a psychotherapeutic treatment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Conners Continuous Performance Test 3rd Edition (CPT 3) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Conners Continuous Performance Test 3rd Edition (CPT 3) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Conners Continuous Performance Test 3rd Edition (CPT 3) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Number subtest of Children's Memory Scale (CMS) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Number subtest of Children's Memory Scale (CMS) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Number subtest of Children's Memory Scale (CMS) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Opposite Worlds subtest of the Test of Everyday Attention for Children (TEA-CH) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A measure of attentional control/switching that requires the child to make cognitive reversals.
Opposite Worlds subtest of the Test of Everyday Attention for Children (TEA-CH) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A measure of attentional control/switching that requires the child to make cognitive reversals.
Opposite Worlds subtest of the Test of Everyday Attention for Children (TEA-CH) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A measure of attentional control/switching that requires the child to make cognitive reversals.
Creature Counting subtest of the Test of Everyday Attention for Children (TEA-CH) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A measure of attentional control and switching that requires children to repeatedly switch between two simple activities, counting upward and counting downward.
Creature Counting subtest of the Test of Everyday Attention for Children (TEA-CH) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A measure of attentional control and switching that requires children to repeatedly switch between two simple activities, counting upward and counting downward.
Creature Counting subtest of the Test of Everyday Attention for Children (TEA-CH) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A measure of attentional control and switching that requires children to repeatedly switch between two simple activities, counting upward and counting downward.
Functional NIRS | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured throughout the training sessions and direct assessments using functional NIRS.
Functional NIRS | Up to 8 to 10 weeks (within the intervention period)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured throughout the training sessions and direct assessments using functional NIRS.
Functional NIRS | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured throughout the training sessions and direct assessments using functional NIRS.
Functional NIRS | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  The levels of oxygenated and deoxygenated hemoglobin of the prefrontal cortex will be measured throughout the training sessions and direct assessments using functional NIRS.

SECONDARY OUTCOMES:
Children's ADHD symptoms | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  Parents and teachers will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.
Children's ADHD symptoms | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Parents and teachers will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.
Children's ADHD symptoms | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents and teachers will be asked to complete the Swanson, Nolan, and Pelham Version IV Scale (SNAP-IV) measuring children's inattentive, hyperactive and impulsive symptoms with a 4-point Likert scale (ranges from 0 to 3). The minimum total score is 0 while the maximum total score is 78, with a higher score indicating a higher level of inattentive, hyperactive and impulsive symptoms.
Behavioural ratings on children's executive functions | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents and teachers will be asked to complete Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation

OTHER OUTCOMES:
Children's enjoyment of the training | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Children's enjoyment of the training will be evaluated using the Cognitive Absorption Scale (CAS) using a 7-point Likert scale (ranges from 1 to 7), which includes four dimensions: temporal dissociation, focused immersion, heightened enjoyment, and curiosity. The total score of this scale ranges from 7 to 119, with a higher score indicating a higher level of children's enjoyment of the training.
Feasibility of conducting VR training within children | Up to 8 to 10 weeks (within the intervention period)
  Children's symptoms of cybersickness (e.g., nausea, fatigue, eye strain) will be measured using the Simulator Sickness Questionnaire (SSQ) after completing every training session, using a 4-point Likert scale (ranges from 0 to 3). The minimum weighted total score of this scale is 0 and the maximum weighted total score is 235.62, with a higher score indicating a higher level of symptoms of cybersickness.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Kar Man SHUM, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be available upon reasonable request. A study protocol of the current study will be available as well.
Supporting Information: Study Protocol
Time Frame: Beginning immediately after publication and ending 5 years after publication.
Access Criteria: To gain access, requestors will need to provide a clear research aim or methodological sound research plan directed to the principal investigator (kkmshum@hku.hk).

REFERENCES:
- [Background] Blume, F., Quixal, M., Hudak, J., Dresler, T., Gawrilow, C., & Ehlis, A. C. (2020). Development of Reading Abilities in Children with ADHD Following fNIRS-Neurofeedback or EMGBiofeedback. Lernen und Lernstörungen, 9(3) 2. Blume, F., Hudak, J., Dresler, T., Ehlis, A. C., Kühnhausen, J., Renner, T. J., & Gawrilow, C. (2017). NIRS-based neurofeedback training in a virtual reality classroom for children with attention-deficit/hyperactivity disorder: study protocol for a randomized controlled trial. Trials, 18(1), 1-16. 3. Marx, A.-M., Ehlis, A.-C., Furdea, A., Holtmann, M., Banaschewski, T., Brandeis, D., … Strehl, U. (2015). Near-infrared spectroscopy (NIRS) neurofeedback as a treatment for children with attention deficit hyperactivity disorder (ADHD): a pilot study. Frontiers in Human Neuroscience, 8(JAN), 1038. 4. Strehl, U., Leins, U., Goth, G., Klinger, C., Hinterberger, T., & Birbaumer, N. (2006). Selfregulation of slow cortical potentials: a new treatment for children with attentiondeficit/hyperactivity disorder. Pediatrics, 118(5), e1530-e1540. 5. Cogmed (2020). Cogmed Working Memory Training. Pearson Clinical Assessment UK. 6. Gau, S. S. F., Lin, C. H., Hu, F. C., Shang, C. Y., Swanson, J. M., Liu, Y. C., & Liu, S. K. (2008). Psychometric properties of the Chinese version of the Swanson, Nolan, and Pelham, version IV scale-Teacher Form. Journal of Pediatric Psychology, 34(8), 850-861. 7. Gau, S. S. F., Shang, C. Y., Liu, S. K., Lin, C. H., Swanson, J. M., Liu, Y. C., & Tu, C. L. (2008). Psychometric properties of the Chinese version of the Swanson, Nolan, and Pelham, version IV scale-parent form. International Journal of Methods in Psychiatric Research, 17(1), 35-44. 8. Gioia, G. A., Isquith, P. K., Guy, S. C., & Kenworthy, L. (2015). BRIEF-2, Behavior Rating Inventory of Executive Function (2nd Ed.). Psychological Assessment Resources, Inc. 9. Shum, K. K. M., Zheng, Q., Chak, G. S., Kei, K. T. L., Lam, C. W. C., Lam, I. K. Y., Lok, C. S. W., & Tang, J. W. Y. (2021). Dimensional structure of the BRIEF2 and its relations with ADHD symptoms and task performance on executive functions in Chinese children. Child Neuropsychology, 27(2), 165-189. 10. Conners, C. K. (2014). Conners Continuous Performance Test 3rd Edition (Conners CPT 3). Multi-Health Systems, Inc. 11. Cohen, M. J. (1997). Children's Memory Scale. The Psychological Corporation. 12. Manly et al. (1998). Test of Everyday Attention for Children. Pearson Clinical Assessment UK. 13. Volpe, R. J., DiPerna, J. C., Hintze, J. M., & Shapiro, E. S. (2005). Observing students in classroom settings: A review of seven coding schemes. School Psychology Review, 34(4), 454-474. 14. Kennedy, R. S., Lane, N. E., Berbaum, K. S., & Lilienthal, M. G. (1993). Simulator sickness questionnaire: An enhanced method for quantifying simulator sickness. The International Journal of Aviation Psychology, 3(3), 203-220. 15. Agarwal, R., & Karahanna, E. (2000). Time flies when you're having fun: Cognitive absorption and beliefs about information technology usage. MIS Quarterly, 24(4), 665-694.
- [Derived] Zheng Q, Kei KT, Chiu KY, Shum KK. Study protocol of a randomised controlled trial of the effects of near-infrared spectroscopy neurofeedback training coupled with virtual reality technology in children with ADHD. BMJ Open. 2024 Dec 7;14(12):e093183. doi: 10.1136/bmjopen-2024-093183. PMID 39645257